CLINICAL TRIAL: NCT06141213
Title: The Relationship Between Fetal Membrane Thickness and Fetal Chromosomal Aneuploidies
Acronym: PLACE2102
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Central Hospital of Gynecology Obstetrics (Other)
Responsible Party: Sponsor
Other Study IDs: PLACE2102
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Chromosome Aberrations
Keywords: Fetal membrane, Fetal chromosomal abnormalities, Ultrasound screening
MeSH Terms: conditions — Chromosome Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal fetal chromosomes: This group will consist of participants with confirmed normal fetal chromosomes.
  Fetal membrane thickness measurements will be taken at enrollment and may be followed up with subsequent measurements throughout the pregnancy.
  The data from this group will serve as the control for comparison with the chromosomal abnormality group.
  Interventions: Diagnostic Test: Ultrasound screening
- Abnormal fetal chromosomes: This group will include participants whose fetuses have been diagnosed with chromosomal abnormalities.
  These participants will also have their fetal membrane thickness measured at the same gestational age as the control group to ensure consistency.
  The comparison of fetal membrane thickness between this group and the control group will be a primary focus of the study.
  Interventions: Diagnostic Test: Ultrasound screening

INTERVENTIONS:
Diagnostic Test: Ultrasound screening — Ultrasound screening for fetal membrane thickness at 18-24 weeks of pregnancy.

SUMMARY:
This observational study aims to recruit pregnant women between 18 to 24 weeks of gestation to investigate the relationship between amniotic membrane thickness and fetal chromosomal abnormalities. The primary objectives are to establish whether a correlation exists between the measured thickness of the amniotic membrane and the presence of chromosomal abnormalities in the fetus, and to determine a cutoff value for amniotic membrane thickness that could indicate an increased risk of such abnormalities. Additionally, the study seeks to assess whether the inclusion of amniotic membrane thickness as a biomarker can enhance the detection rate of non-invasive prenatal testing (NIPT) and nuchal translucency (NT) for chromosomal abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnant women between 18-24 weeks of gestation.
2. Participants with high-risk indications for prenatal fetal chromosomal abnormalities, including:

   * Nuchal translucency (NT) ≥ 3 mm.
   * High-risk results from non-invasive prenatal testing (NIPT) using cell-free fetal DNA from peripheral maternal blood.
   * Ultrasound-detected fetal abnormalities.
   * Other indicators include adverse birth histories, parental chromosomal abnormalities, familial diseases, and a history of thyroid cancer post-surgery.
3. Gestational age and estimated due date were confirmed by the first day of the last menstrual period and adjusted using fetal crown-rump length measured during the first-trimester ultrasound scan.
4. Participants who provided written informed consent for amniocentesis.

   -

Exclusion Criteria:

1. Women with multiple pregnancies or higher-order births.
2. Previous chorionic villus sampling or amniocentesis in the current pregnancy.
3. Gestational age at the time of amniocentesis greater than 25 weeks or less than 18 weeks.
4. Presence of amniotic band syndrome.
5. The presence of uterine anomalies or conditions may impact ultrasound measurements' reliability.
6. Any medical condition or obstetric complication that, in the opinion of the investigators, might pose a risk to the participant or interfere with the study outcomes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population included pregnant women referred to the Center for Prenatal Diagnosis and Fetal Medicine at Tianjin Central Hospital of Obstetrics and Gynecology. These participants were identified based on clinical indicators of elevated risk for fetal chromosomal abnormalities. The cohort represented a diverse age range of expectant mothers, predominantly from Tianjin's urban and suburban regions in China.
  Focused on singleton pregnancies, the study minimizes variables linked to the complexities of multiple gestations. The women were chiefly in their second trimester, a pivotal time for fetal development and diagnostic evaluation.
  A considerable portion of the study participants had received high-risk NIPT results or demonstrated ultrasound markers suggesting potential chromosomal irregularities. This selection was vital for evaluating FM thickness as a diagnostic tool for chromosomal anomalies.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Fetal Membrane Thickness and Chromosomal Abnormalities | March, 2024
  The difference in mean fetal membrane thickness between the normal and abnormal chromosomal groups, and the establishment of a threshold value for risk assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Central Hospital of Obstetrics and Gynecology, Tianjin, Tianjin Municipality, China